CLINICAL TRIAL: NCT03332706
Title: Department of Gynecology and Obstetrics From Peking Union Medical College Hospital
Brief Title: the Association Between Blood's and Urinary Heavy Metal Level in Pregnant Women and the Spontaneous Abortion
Acronym: HMLandSA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HML2017
Record Dates: First submitted 2017-11-02; First posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Heavy Metal Toxicity; Spontaneous Abortion
MeSH Terms: conditions — Heavy Metal Poisoning; Abortion, Spontaneous | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SG: Study Group is the group where the patients during observation suffer from spontaneous abortion or missed abortion,
  Interventions: Other: observation
- CG: Control Group is where the patients carry the normal live fetal for at least 8 weeks
  Interventions: Other: observation

INTERVENTIONS:
Other: observation — after the subjects are included into the groups,they are asked to do a questionaire.Then,we just observe the outcomes of pregnancy

SUMMARY:
The aim of the study was to define the possible association between heavy iron level and the consequence of pregnancy especially spontaneous abortion and missed abortion. The study population will comprised the first-trimester pregnant women in the PUMCH (Peking Union Medicine College Hospital) during 2017 October to 2018 November. We categorised the patients into two groups, the study group where the patients suffered from spontaneous abortion or missed abortion, and the control group where the patients carry the normal live fetal for at least 8 weeks and ask for artificial abortion. All the cases included in the study were examined with respect to 6 kinds of heavy iron level in venous blood and urine, then correlation analysis was applied to define heavy iron level between two groups.

ELIGIBILITY:
Inclusion Criteria:

- early trimester pregnant women

Exclusion Criteria:

-

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: the first-trimester pregnant women in the PUMCH (Peking Union Medicine College Hospital) during 2017 October to 2018 November.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-10-10 (Actual); Primary Completion 2018-11-01 (Estimated); Study Completion 2018-11-30 (Estimated)

PRIMARY OUTCOMES:
blood's and urinary heavy metal level | 12months
  6 kinds of heavy metal:Pb,As,Hg,Gd,Cr,Se

CONTACTS AND LOCATIONS:
Overall Officials: Liu xinyan, Study Director — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Pekin, China

IPD SHARING:
Plan to Share IPD: Undecided